CLINICAL TRIAL: NCT04625647
Title: A Phase II Study of AMG 510 in Participants With Previously Treated Stage IV or Recurrent KRAS G12C Mutated Non-Squamous Non-Small Cell Lung Cancer (ECOG-ACRIN LUNG-MAP SUB-STUDY)
Brief Title: Testing the Use of Targeted Treatment (AMG 510) for KRAS G12C Mutated Advanced Non-squamous Non-small Cell Lung Cancer (A Lung-MAP Treatment Trial)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S1900E; NCI-2020-08103 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); S1900E (Other: SWOG); S1900E (Other: CTEP); U10CA180888 (NIH)
Record Dates: First submitted 2020-11-06; First posted 2020-11-12 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Lung Adenocarcinoma; Lung Non-Small Cell Carcinoma; Recurrent Lung Non-Squamous Non-Small Cell Carcinoma; Stage IV Lung Cancer AJCC v8; Stage IVA Lung Cancer AJCC v8; Stage IVB Lung Cancer AJCC v8
MeSH Terms: conditions — Adenocarcinoma of Lung; Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — sotorasib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (AMG 510) (Experimental): Patients receive AMG 510 PO QD on days 1-21. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Sotorasib

INTERVENTIONS:
Drug: Sotorasib — Given PO
  Other Names: AMG 510; AMG-510; AMG510

SUMMARY:
This phase II Lung-MAP treatment trial studies the effect of AMG 510 in treating non-squamous non-small cell lung cancer that is stage IV or has come back (recurrent) and has a specific mutation in the KRAS gene, known as KRAS G12C. Mutations in this gene may cause the cancer to grow. AMG 510, a targeted treatment against the KRAS G12C mutation, may help stop the growth of tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the response rate (confirmed, complete or partial) of AMG 510 in participants with KRAS^G12C mutated stage IV or recurrent non-squamous non-small cell lung cancer (NSCLC).

SECONDARY OBJECTIVES:

I. To evaluate investigator assessed progression-free survival (IA-PFS) within each cohort.

II. To evaluate overall survival (OS) within each cohort. III. To evaluate duration of response (DOR) among responders within each cohort.

IV. To evaluate the frequency and severity of toxicities within the full study population (all cohorts combined).

TRANSLATIONAL MEDICINE OBJECTIVES:

I. To evaluate the association between clinical outcomes (response, IA-PFS, OS) and other co-mutations (e.g., CDKN2A/B/C, ATM, PIK3CA) identified by the Foundation Medicine Inc (FMI) FoundationOne CDx from LUNGMAP, within cohorts and across the full study population of KRAS^G12C positive participants.

II. To evaluate the association between clinical outcomes (response, IA-PFS, OS) and PD-L1 total proportion score determined by screening in LUNGMAP, within cohorts and across the full study population of KRAS^G12C positive participants.

III. To evaluate the association between clinical outcomes (response, IA-PFS, OS) and Tumor Mutational Burden Score determined by the FMI FoundationOne CDx from LUNGMAP, within cohorts and across the full study population of KRAS^G12C positive participants.

IV. To collect, process, and bank cell-free deoxyribonucleic acid (cfDNA) at pre-treatment on cycle 1 day 1, cycle 2 day 1, cycle 3 day 1, and at progression for future development of a proposal to evaluate comprehensive next-generation sequencing of circulating tumor DNA (ctDNA) and association with clinical outcomes.

Note: The translational medicine proposal to use these specimens will be submitted as a revision to CTEP for approval, prior to the SWOG Statistical and Data Management Center (SDMC) review of assay results.

OUTLINE:

Patients receive AMG 510 orally (PO) once daily (QD) on days 1-21. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 3 years if the disease has not gotten worse at the time of finishing study treatment. If the disease has gotten worse, patients are followed up every 6 months for 2 years, then at the end of the 3 years from the time they go on study.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be assigned to S1900E. Assignment to S1900E is determined by the LUNGMAP protocol genomic profiling using the FoundationOne assay. Biomarker eligibility for S1900E is based on the identification of a KRAS^G12C mutation
* Participants must have confirmed stage IV or recurrent non-squamous non-small cell lung cancer (NSCLC). Mixed histology NSCLC with less than 50% squamous component is allowed
* Participants must have measurable disease documented by computed tomography (CT) or magnetic resonance imaging (MRI). The CT from a combined positron emission tomography (PET)/CT may be used to document only non-measurable disease unless it is of diagnostic quality. Measurable disease must be assessed within 28 days prior to sub-study registration. Pleural effusions, ascites and laboratory parameters are not acceptable as the only evidence of disease. Non-measurable disease must be assessed within 42 days prior to sub-study registration. Participants whose only measurable disease is within a previous radiation therapy port must demonstrate clearly progressive disease (in the opinion of the treating investigator) prior to registration
* Participants must have a CT or MRI scan of the brain to evaluate for central nervous system (CNS) disease within 42 days prior to sub-study registration
* Participants with known human immunodeficiency virus (HIV) infection must be receiving anti-retroviral therapy and have an undetectable viral load at their most recent viral load test within 6 months prior to sub-study registration
* Participants with EGFR sensitizing mutations, EGFR T790M mutation, ALK gene fusion, ROS1 gene rearrangement, or BRAF V600E mutation must have progressed following all standard of care targeted therapy
* Participants with spinal cord compression or brain metastases must have received local treatment to these metastases and remained clinically controlled and asymptomatic for at least 7 days following stereotactic radiation and/or 14 days following whole brain radiation, and prior to sub-study registration
* Participants must have received at least one line of systemic treatment for stage IV or recurrent NSCLC
* Participants must have progressed (in the opinion of the treating physician) following the most recent line of systemic therapy for NSCLC
* Participants must have recovered (=< grade 1) from side effects of prior therapy. The exception is if a side effect from a prior treatment is known to be permanent without expected further recovery or resolution (i.e., endocrinopathy from immunotherapy or cisplatin neurotoxicity)
* Participants must be able to swallow tablets whole
* Pre-study history and physical exam must be obtained within 28 days prior to sub-study registration
* Absolute neutrophil count (ANC) >= 1,500/uL obtained within 28 days prior to sub-study registration
* Platelet count >= 75,000/uL obtained within 28 days prior to sub-study registration
* Hemoglobin >= 9 g/dL obtained within 28 days prior to sub-study registration
* Serum bilirubin =< institutional upper limit of normal (IULN) within 28 days prior to sub-study registration
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 2 x IULN within 28 days prior to sub-study registration. For participants with liver metastases, and ALT and AST must be =< 5 x IULN
* Participants must have a serum creatinine =< 1.5 x IULN or calculated creatinine clearance >= 50 mL/min using the following Cockcroft-Gault Formula. This specimen must have been drawn and processed within 28 days prior to sub-study registration
* Participants must have Zubrod performance status 0-1 documented within 28 days prior to sub-study registration
* Participants of reproductive potential must have a negative serum pregnancy test within 28 days prior to sub-study registration
* Participants must agree to have blood specimens submitted for circulating tumor DNA (ctDNA)
* Participants must be offered the opportunity to participate in specimen banking and in correlative studies for collection and future use of specimens. With participant consent, specimens must be collected and submitted via the Southwest Oncology Group (SWOG) Specimen Tracking System
* Participants must be informed of the investigational nature of this study and must sign and give informed consent in accordance with institutional and federal guidelines

  * NOTE: As a part of the Oncology Patient Enrollment Network (OPEN) registration process the treating institution's identity is provided in order to ensure that the current (within 365 days) date of institutional review board approval for this study has been entered in the system
* As a part of the Oncology Patient Enrollment Network (OPEN) registration process the treating institution's identity is provided in order to ensure that the current (within 365 days) date of institutional review board approval for this study has been entered in the system
* Participants with impaired decision-making capacity are eligible as long as their neurological or psychological condition does not preclude their safe participation in the study (e.g., tracking pill consumption and reporting adverse events to the investigator). For participants with impaired decision-making capabilities, legally authorized representatives may sign and give informed consent on behalf of study participants in accordance with applicable federal, local, and Central Institutional Review Board (CIRB) regulations

Exclusion Criteria:

* Participants with spinal cord compression or brain metastases must not have residual neurological dysfunction, unless no further recovery is expected, and the participant has been stable on weaning doses of corticosteroids prior to sub-study registration
* Participants must not have leptomeningeal disease unless: (1) asymptomatic and (2) only detected on radiographic imaging (i.e., not present in cytology from cerebral spinal fluid [CSF] if CSF sampled)
* Participants must not have received any prior systemic therapy (systemic chemotherapy, immunotherapy or investigational drug) within 21 days prior to sub-study registration
* Participants must not have received any radiation therapy within 14 days prior to sub-study registration, with the exception of stereotactic radiation to CNS metastases which must have been completed at least 7 days prior to sub-study registration
* Participants must not have received prior AMG 510 or other KRAS^G12C specific inhibitor
* Participants must not be planning to receive any concurrent chemotherapy, immunotherapy, biologic or hormonal therapy for cancer treatment while receiving treatment on this study
* Participants must not have had a major surgery within 14 days prior to sub-study registration. Participant must have fully recovered from the effects of prior surgery in the opinion of the treating investigator
* Participants must not have any grade III/IV cardiac disease as defined by the New York Heart Association criteria (i.e., participants with cardiac disease resulting in marked limitation of physical activity or resulting in inability to carry on any physical activity without discomfort), unstable angina pectoris, and myocardial infarction within 6 months, or serious uncontrolled cardiac arrhythmia
* Participants must not have a prior or concurrent malignancy whose natural history or treatment has the potential to interfere with the safety or efficacy assessment of the investigational regimen
* Participants must not have gastrointestinal disorders that may impact drug absorption
* Participants must not have received strong inducers of CYP3A4 (including herbal supplements such as St. John's wort) within 14 days prior to sub-study registration and must not be planning to use strong inducers of CYP3A4 throughout protocol treatment
* Participants must not have received CYP3A4 sensitive substrates (with a narrow therapeutic window) within 14 days prior to sub-study registration and must not be planning to use CYP3A4 sensitive substrates (with a narrow therapeutic window) throughout protocol treatment
* Participants must not be pregnant or nursing. Participants with uteri must have agreed to use an effective contraceptive method for at least one month after the last dose of AMG 510. Participants with sperm must have agreed to use an effective contraceptive method for at least 3 months after the last dose of AMG 510. Participants are considered to be of "reproductive potential" if they have had menses at any time in the preceding 12 consecutive months and no prior oophorectomy and/or hysterectomy. In addition to routine contraceptive methods, "effective contraception" for participants with uteri also includes heterosexual celibacy and surgery intended to prevent pregnancy (or with a side-effect of pregnancy prevention) defined as a hysterectomy, bilateral oophorectomy or bilateral tubal ligation. Acceptable methods of birth control for participants with sperm include sexual abstinence (refraining from heterosexual intercourse); vasectomy with testing showing there is no sperm in the semen; bilateral tubal ligation or occlusion in the partner; or a condom (the female partner should also consider a form of birth control). However, if at any point a previously celibate participant chooses to become heterosexually active during the time period for use of contraceptive measures outlined in the protocol, he/she is responsible for beginning contraceptive measures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2021-04-16 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Response rate (confirmed, complete or partial) | Up to 3 years

SECONDARY OUTCOMES:
Incidence of adverse events | Up to 3 years
  The frequency and grade of individual toxicities attributable to treatment will be estimated.
Progression free survival | Up to 3 years
  Will be estimated using the method of Kaplan-Meier. Confidence intervals about medians will be estimated using the Brookmeyer-Crowley method and about landmark time points will be calculated using Greenwood's formula and based on a log-log transformation applied on the survival function. Binary proportions and associated confidence intervals will be estimated for within cohort objectives. With participants in Cohort 1 and 3 and participants in Cohort 2, binary proportions can be estimated to within 16% and 20% with 95% confidence, respectively.
Overall survival | Up to 3 years
  Will be estimated using the method of Kaplan-Meier. Confidence intervals about medians will be estimated using the Brookmeyer-Crowley method and about landmark time points will be calculated using Greenwood's formula and based on a log-log transformation applied on the survival function. Binary proportions and associated confidence intervals will be estimated for within cohort objectives. With participants in Cohort 1 and 3 and participants in Cohort 2, binary proportions can be estimated to within 16% and 20% with 95% confidence, respectively.
Duration of response | Up to 3 years
  Will be estimated using the method of Kaplan-Meier. Confidence intervals about medians will be estimated using the Brookmeyer-Crowley method and about landmark time points will be calculated using Greenwood's formula and based on a log-log transformation applied on the survival function. Binary proportions and associated confidence intervals will be estimated for within cohort objectives. With participants in Cohort 1 and 3 and participants in Cohort 2, binary proportions can be estimated to within 16% and 20% with 95% confidence, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Sukhmani K Padda, Principal Investigator — SWOG Cancer Research Network
Locations (829):
- United States (828):
  - Veterans Administration Medical Center - Birmingham, Birmingham, Alabama
  - Anchorage Associates in Radiation Medicine, Anchorage, Alaska
  - Anchorage Radiation Therapy Center, Anchorage, Alaska
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Fairbanks Memorial Hospital, Fairbanks, Alaska
  - Kingman Regional Medical Center, Kingman, Arizona
  - Cancer Center at Saint Joseph's, Phoenix, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - Mercy Hospital Fort Smith, Fort Smith, Arkansas
  - CHI Saint Vincent Cancer Center Hot Springs, Hot Springs, Arkansas
  - NEA Baptist Memorial Hospital and Fowler Family Cancer Center - Jonesboro, Jonesboro, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Kaiser Permanente-Anaheim, Anaheim, California
  - Mission Hope Medical Oncology - Arroyo Grande, Arroyo Grande, California
  - PCR Oncology, Arroyo Grande, California
  - Sutter Auburn Faith Hospital, Auburn, California
  - Sutter Cancer Centers Radiation Oncology Services-Auburn, Auburn, California
  - Kaiser Permanente-Baldwin Park, Baldwin Park, California
  - Kaiser Permanente-Bellflower, Bellflower, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Tower Cancer Research Foundation, Beverly Hills, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Sutter Cancer Centers Radiation Oncology Services-Cameron Park, Cameron Park, California
  - Eden Hospital Medical Center, Castro Valley, California
  - Sutter Davis Hospital, Davis, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Kaiser Permanente-Fontana, Fontana, California
  - Palo Alto Medical Foundation-Fremont, Fremont, California
  - Kaiser Permanente-Fresno, Fresno, California
  - Kaiser Permanente South Bay, Harbor City, California
  - Kaiser Permanente-Irvine, Irvine, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Tibor Rubin VA Medical Center, Long Beach, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Kaiser Permanente West Los Angeles, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Fremont - Rideout Cancer Center, Marysville, California
  - Memorial Medical Center, Modesto, California
  - Palo Alto Medical Foundation-Camino Division, Mountain View, California
  - Palo Alto Medical Foundation-Gynecologic Oncology, Mountain View, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Kaiser Permanente-Ontario, Ontario, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - Kaiser Permanente - Panorama City, Panorama City, California
  - Eisenhower Medical Center, Rancho Mirage, California
  - Kaiser Permanente-Riverside, Riverside, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Sutter Cancer Centers Radiation Oncology Services-Roseville, Roseville, California
  - Sutter Roseville Medical Center, Roseville, California
  - Kaiser Permanente Downtown Commons, Sacramento, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Kaiser Permanente-San Diego Mission, San Diego, California
  - Kaiser Permanente-San Diego Zion, San Diego, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - Veterans Affairs Medical Center - San Francisco, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Pacific Central Coast Health Center-San Luis Obispo, San Luis Obispo, California
  - Kaiser Permanente-San Marcos, San Marcos, California
  - Mills Health Center, San Mateo, California
  - Kaiser San Rafael-Gallinas, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Palo Alto Medical Foundation-Santa Cruz, Santa Cruz, California
  - Mission Hope Medical Oncology - Santa Maria, Santa Maria, California
  - Sutter Pacific Medical Foundation, Santa Rosa, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Saint Helena Hospital, St. Helena, California
  - Palo Alto Medical Foundation-Sunnyvale, Sunnyvale, California
  - Cedars-Sinai Cancer - Tarzana, Tarzana, California
  - Torrance Memorial Physician Network - Cancer Care, Torrance, California
  - Gene Upshaw Memorial Tahoe Forest Cancer Center, Truckee, California
  - City of Hope Upland, Upland, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - Presbyterian Intercommunity Hospital, Whittier, California
  - Kaiser Permanente-Woodland Hills, Woodland Hills, California
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - The Medical Center of Aurora, Aurora, Colorado
  - Boulder Community Foothills Hospital, Boulder, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Rocky Mountain Cancer Centers - Centennial, Centennial, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - The Women's Imaging Center, Denver, Colorado
  - AdventHealth Porter, Denver, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Western Surgical Care, Denver, Colorado
  - CommonSpirit Cancer Center Mercy, Durango, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Mountain Blue Cancer Care Center - Swedish, Englewood, Colorado
  - Rocky Mountain Cancer Centers - Swedish, Englewood, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - The Melanoma and Skin Cancer Institute, Englewood, Colorado
  - Banner North Colorado Medical Center, Greeley, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - AdventHealth Littleton, Littleton, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - Banner North Colorado Medical Center - Loveland Campus, Loveland, Colorado
  - AdventHealth Parker, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Rocky Mountain Cancer Centers-Thornton, Thornton, Colorado
  - Smilow Cancer Hospital-Derby Care Center, Derby, Connecticut
  - Smilow Cancer Hospital Care Center-Fairfield, Fairfield, Connecticut
  - Smilow Cancer Hospital Care Center at Glastonbury, Glastonbury, Connecticut
  - Smilow Cancer Hospital Care Center at Greenwich, Greenwich, Connecticut
  - Smilow Cancer Hospital Care Center - Guilford, Guilford, Connecticut
  - Hartford Hospital, Hartford, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Midstate Medical Center, Meriden, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Yale University, New Haven, Connecticut
  - Yale-New Haven Hospital North Haven Medical Center, North Haven, Connecticut
  - Smilow Cancer Hospital-Orange Care Center, Orange, Connecticut
  - Smilow Cancer Hospital Care Center at Long Ridge, Stamford, Connecticut
  - Smilow Cancer Hospital-Torrington Care Center, Torrington, Connecticut
  - Smilow Cancer Hospital Care Center-Trumbull, Trumbull, Connecticut
  - Smilow Cancer Hospital-Waterbury Care Center, Waterbury, Connecticut
  - Smilow Cancer Hospital Care Center - Waterford, Waterford, Connecticut
  - Veterans Affairs Connecticut Healthcare System-West Haven Campus, West Haven, Connecticut
  - Bayhealth Hospital Kent Campus, Dover, Delaware
  - Beebe Medical Center, Lewes, Delaware
  - Bayhealth Hospital Sussex Campus, Milford, Delaware
  - Beebe South Coastal Health Campus, Millville, Delaware
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - TidalHealth Nanticoke / Allen Cancer Center, Seaford, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - Kaiser Permanente-Capitol Hill Medical Center, Washington D.C., District of Columbia
  - Mount Sinai Comprehensive Cancer Center at Aventura, Aventura, Florida
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Moffitt Cancer Center-International Plaza, Tampa, Florida
  - Moffitt Cancer Center - McKinley Campus, Tampa, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Cleveland Clinic-Weston, Weston, Florida
  - Northside Hospital, Atlanta, Georgia
  - Northeast Georgia Medical Center Braselton, Braselton, Georgia
  - Atlanta VA Medical Center, Decatur, Georgia
  - Northside Hospital - Duluth, Duluth, Georgia
  - Northeast Georgia Medical Center-Gainesville, Gainesville, Georgia
  - Northside Hospital - Gwinnett, Lawrenceville, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Suburban Hematology Oncology Associates - Snellville, Snellville, Georgia
  - South Georgia Medical Center/Pearlman Cancer Center, Valdosta, Georgia
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Queen's Cancer Cenrer - POB I, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Hawaii Cancer Care Inc-Liliha, Honolulu, Hawaii
  - Hawaii Diagnostic Radiology Services LLC, Honolulu, Hawaii
  - Kuakini Medical Center, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Straub Medical Center - Kahului Clinic, Kahului, Hawaii
  - Castle Medical Center, Kailua, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Hawaii Cancer Care - Westridge, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Queen's Cancer Center - Pearlridge, ‘Aiea, Hawaii
  - The Cancer Center of Hawaii-Pali Momi, ‘Aiea, Hawaii
  - The Queen's Medical Center - West Oahu, ‘Ewa Beach, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Walter Knox Memorial Hospital, Emmett, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - OSF Saint Anthony's Health Center, Alton, Illinois
  - Rush-Copley Medical Center, Aurora, Illinois
  - Advocate Good Shepherd Hospital, Barrington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Advocate Illinois Masonic Medical Center, Chicago, Illinois
  - AMG Crystal Lake - Oncology, Crystal Lake, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Illinois CancerCare-Dixon, Dixon, Illinois
  - Advocate Good Samaritan Hospital, Downers Grove, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Advocate Sherman Hospital, Elgin, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - NorthShore University HealthSystem-Glenbrook Hospital, Glenview, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Advocate South Suburban Hospital, Hazel Crest, Illinois
  - NorthShore University HealthSystem-Highland Park Hospital, Highland Park, Illinois
  - Edward Hines Jr VA Hospital, Hines, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - AMG Libertyville - Oncology, Libertyville, Illinois
  - Condell Memorial Hospital, Libertyville, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - SSM Health Good Samaritan, Mount Vernon, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - OSF Saint Anthony Medical Center, Rockford, Illinois
  - MercyOne Genesis Silvis Cancer Center, Silvis, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Illinois CancerCare - Washington, Washington, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Parkview Regional Medical Center, Fort Wayne, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Richard L. Roudebush Veterans Affairs Medical Center, Indianapolis, Indiana
  - Franciscan Health Indianapolis, Indianapolis, Indiana
  - Woodland Cancer Care Center, Michigan City, Indiana
  - Franciscan Health Mooresville, Mooresville, Indiana
  - Reid Health, Richmond, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Union Hospital, Terre Haute, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic - Ames, Ames, Iowa
  - UI Health Care Mission Cancer and Blood - Ankeny Clinic, Ankeny, Iowa
  - McFarland Clinic - Boone, Boone, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Alegent Health Mercy Hospital, Council Bluffs, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - MercyOne Genesis Davenport Medical Center, Davenport, Iowa
  - MercyOne Genesis Davenport Cancer Center, Davenport, Iowa
  - Iowa Cancer Specialists, Davenport, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - McFarland Clinic - Trinity Cancer Center, Fort Dodge, Iowa
  - McFarland Clinic - Jefferson, Jefferson, Iowa
  - McFarland Clinic - Marshalltown, Marshalltown, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Central Care Cancer Center - Garden City, Garden City, Kansas
  - Central Care Cancer Center - Great Bend, Great Bend, Kansas
  - HaysMed, Hays, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - The University of Kansas Cancer Center - Olathe, Olathe, Kansas
  - Freeman Physician Group of Pittsburg, Pittsburg, Kansas
  - Mercy Hospital Pittsburg, Pittsburg, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - Cotton O'Neil Cancer Center / Stormont Vail Health, Topeka, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Baptist Health Corbin, Corbin, Kentucky
  - Commonwealth Cancer Center-Corbin, Corbin, Kentucky
  - Baptist Health Lexington, Lexington, Kentucky
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Baptist Health Hamburg, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Saint Joseph London, London, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - Baptist Health Louisville, Louisville, Kentucky
  - Saints Mary and Elizabeth Hospital, Louisville, Kentucky
  - UofL Health Medical Center Northeast, Louisville, Kentucky
  - Jewish Hospital Medical Center South, Shepherdsville, Kentucky
  - Medical Center of Baton Rouge, Baton Rouge, Louisiana
  - Ochsner High Grove, Baton Rouge, Louisiana
  - Ochsner Medical Center Kenner, Kenner, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Lafayette Family Cancer Center-EMMC, Brewer, Maine
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Saint Agnes Hospital, Baltimore, Maryland
  - Kaiser Permanente-Woodlawn Medical Center, Baltimore, Maryland
  - UPMC Western Maryland, Cumberland, Maryland
  - Kaiser Permanente-Gaithersburg Medical Center, Gaithersburg, Maryland
  - Kaiser Permanente - Largo Medical Center, Largo, Maryland
  - Kaiser Permanente Lutherville - Timonium Medical Center, Lutherville, Maryland
  - Beverly Hospital, Beverly, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Addison Gilbert Hospital, Gloucester, Massachusetts
  - Boston Veteran's Affairs Medical Center, Jamaica Plain, Massachusetts
  - Lahey Medical Center-Peabody, Peabody, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - UMass Memorial Medical Center - University Campus, Worcester, Massachusetts
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Trinity Health Medical Center - Brighton, Brighton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health Medical Center - Canton, Canton, Michigan
  - Caro Cancer Center, Caro, Michigan
  - Chelsea Hospital, Chelsea, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Hematology Oncology Consultants-Clarkston, Clarkston, Michigan
  - Newland Medical Associates-Clarkston, Clarkston, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - Henry Ford River District Hospital, East China Township, Michigan
  - Cancer Hematology Centers - Flint, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - Henry Ford Saint John Hospital - Academic, Grosse Pointe Woods, Michigan
  - Henry Ford Saint John Hospital - Breast, Grosse Pointe Woods, Michigan
  - Henry Ford Saint John Hospital - Van Elslander, Grosse Pointe Woods, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Beacon Kalamazoo Cancer Center, Kalamazoo, Michigan
  - Beacon Kalamazoo, Kalamazoo, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Hope Cancer Clinic, Livonia, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Henry Ford Saint John Hospital - Macomb Medical, Macomb, Michigan
  - Henry Ford Warren Hospital - Breast Macomb, Macomb, Michigan
  - Saint Mary's Oncology/Hematology Associates of Marlette, Marlette, Michigan
  - Trinity Health Muskegon Hospital, Muskegon, Michigan
  - Corewell Health Lakeland Hospitals - Niles Hospital, Niles, Michigan
  - Cancer and Hematology Centers of Western Michigan - Norton Shores, Norton Shores, Michigan
  - Hope Cancer Center, Pontiac, Michigan
  - Michigan Healthcare Professionals Pontiac, Pontiac, Michigan
  - Newland Medical Associates-Pontiac, Pontiac, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Corewell Health Reed City Hospital, Reed City, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Oncology Hematology Associates of Saginaw Valley PC, Saginaw, Michigan
  - Corewell Health Lakeland Hospitals - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Corewell Health Lakeland Hospitals - Saint Joseph Hospital, Saint Joseph, Michigan
  - Bhadresh Nayak MD PC-Sterling Heights, Sterling Heights, Michigan
  - MyMichigan Medical Center Tawas, Tawas City, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Advanced Breast Care Center PLLC, Warren, Michigan
  - Henry Ford Health Warren Hospital, Warren, Michigan
  - Henry Ford Madison Heights Hospital - Breast, Warren, Michigan
  - Henry Ford Warren Hospital - GLCMS, Warren, Michigan
  - Macomb Hematology Oncology PC, Warren, Michigan
  - Saint Mary's Oncology/Hematology Associates of West Branch, West Branch, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Huron Gastroenterology PC, Ypsilanti, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Riverwood Healthcare Center, Aitkin, Minnesota
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Minnesota Oncology - Burnsville, Burnsville, Minnesota
  - Cambridge Medical Center, Cambridge, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health - Deer River Clinic, Deer River, Minnesota
  - Essentia Health Saint Mary's - Detroit Lakes Clinic, Detroit Lakes, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Lake Region Healthcare Corporation-Cancer Care, Fergus Falls, Minnesota
  - Essentia Health - Fosston, Fosston, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Minneapolis VA Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - Monticello Cancer Center, Monticello, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - Essentia Health - Park Rapids, Park Rapids, Minnesota
  - Fairview Northland Medical Center, Princeton, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Essentia Health Sandstone, Sandstone, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Sanford Thief River Falls Medical Center, Thief River Falls, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Sanford Cancer Center Worthington, Worthington, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - Baptist Memorial Hospital and Cancer Center-Golden Triangle, Columbus, Mississippi
  - Baptist Cancer Center-Grenada, Grenada, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Union County, New Albany, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Oxford, Oxford, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Desoto, Southhaven, Mississippi
  - Mercy Oncology and Hematology - Clayton-Clarkson, Ballwin, Missouri
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Mercy Cancer Center - Cape Girardeau, Cape Girardeau, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - MU Health Care Goldschmidt Cancer Center, Jefferson City, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - University Health Truman Medical Center, Kansas City, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Phelps Health Delbert Day Cancer Institute, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Mercy Infusion Center - Chippewa, St Louis, Missouri
  - Veteran's Affairs Medical Center - Saint Louis, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Mercy Hospital Washington, Washington, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Center, Missoula, Montana
  - Nebraska Cancer Specialists/Oncology Hematology West PC, Grand Island, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Saint Elizabeth Regional Medical Center, Lincoln, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Midlands Community Hospital, Papillion, Nebraska
  - Carson Tahoe Regional Medical Center, Carson City, Nevada
  - Cancer and Blood Specialists-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Horizon Ridge, Henderson, Nevada
  - Las Vegas Cancer Center-Henderson, Henderson, Nevada
  - OptumCare Cancer Care at Seven Hills, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Southeast Henderson, Henderson, Nevada
  - Las Vegas Urology - Green Valley, Henderson, Nevada
  - Las Vegas Urology - Pebble, Henderson, Nevada
  - Oncology Las Vegas - Henderson, Henderson, Nevada
  - Urology Specialists of Nevada - Green Valley, Henderson, Nevada
  - Las Vegas Urology - Pecos, Las Vegas, Nevada
  - Desert West Surgery, Las Vegas, Nevada
  - OptumCare Cancer Care at Charleston, Las Vegas, Nevada
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Hope Cancer Care of Nevada, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - Urology Specialists of Nevada - Central, Las Vegas, Nevada
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - Las Vegas Prostate Cancer Center, Las Vegas, Nevada
  - Las Vegas Urology - Sunset, Las Vegas, Nevada
  - Urology Specialists of Nevada - Southwest, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - Ann M Wierman MD LTD, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - Las Vegas Urology - Cathedral Rock, Las Vegas, Nevada
  - Las Vegas Urology - Smoke Ranch, Las Vegas, Nevada
  - Oncology Las Vegas - Tenaya, Las Vegas, Nevada
  - OptumCare Cancer Care at MountainView, Las Vegas, Nevada
  - Urology Specialists of Nevada - Northwest, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Town Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Las Vegas Cancer Center-Medical Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - University Cancer Center, Las Vegas, Nevada
  - Hope Cancer Care of Nevada-Pahrump, Pahrump, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Saint Mary's Regional Medical Center, Reno, Nevada
  - Radiation Oncology Associates, Reno, Nevada
  - New Hampshire Oncology Hematology PA-Concord, Concord, New Hampshire
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Solinsky Center for Cancer Care, Manchester, New Hampshire
  - Ocean University Medical Center, Brick, New Jersey
  - Southern Ocean County Medical Center, Manahawkin, New Jersey
  - Virtua Samson Cancer Center, Moorestown, New Jersey
  - Virtua Memorial, Mount Holly, New Jersey
  - Jersey Shore Medical Center, Neptune City, New Jersey
  - Riverview Medical Center/Booker Cancer Center, Red Bank, New Jersey
  - Virtua Voorhees, Voorhees Township, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Presbyterian Kaseman Hospital, Albuquerque, New Mexico
  - Presbyterian Rust Medical Center/Jorgensen Cancer Center, Rio Rancho, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - Mary Imogene Bassett Hospital, Cooperstown, New York
  - The Cancer Institute at Saint Francis Hospital, East Hills, New York
  - Arnot Ogden Medical Center/Falck Cancer Center, Elmira, New York
  - Glens Falls Hospital, Glens Falls, New York
  - University of Rochester, Rochester, New York
  - James J Peters VA Medical Center, The Bronx, New York
  - Good Samaritan University Hospital, West Islip, New York
  - Cone Health Cancer Center at Asheboro, Asheboro, North Carolina
  - Randolph Hospital, Asheboro, North Carolina
  - Cone Health MedCenter Asheboro, Asheboro, North Carolina
  - AdventHealth Infusion Center Asheville, Asheville, North Carolina
  - Cone Health Cancer Center at Alamance Regional, Burlington, North Carolina
  - AdventHealth Infusion Center Haywood, Clyde, North Carolina
  - Durham VA Medical Center, Durham, North Carolina
  - Cone Health Cancer Center, Greensboro, North Carolina
  - Cone Health Cancer Center at Drawbridge Parkway, Greensboro, North Carolina
  - AdventHealth Hendersonville, Hendersonville, North Carolina
  - Cone Heath Cancer Center at Mebane, Mebane, North Carolina
  - Annie Penn Memorial Hospital, Reidsville, North Carolina
  - AdventHealth Infusion Center Weaverville, Weaverville, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Essentia Health Cancer Center-South University Clinic, Fargo, North Dakota
  - Sanford South University Medical Center, Fargo, North Dakota
  - Southpointe-Sanford Medical Center Fargo, Fargo, North Dakota
  - Sanford Medical Center Fargo, Fargo, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Essentia Health - Jamestown Clinic, Jamestown, North Dakota
  - Aultman Alliance Community Hospital, Alliance, Ohio
  - Indu and Raj Soin Medical Center, Beavercreek, Ohio
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Saint Elizabeth Boardman Hospital, Boardman, Ohio
  - Cleveland Clinic Mercy Hospital, Canton, Ohio
  - Aultman Health Foundation, Canton, Ohio
  - Dayton Physicians LLC-Miami Valley South, Centerville, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Kenwood, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - TriHealth Cancer Institute-Westside, Cincinnati, Ohio
  - TriHealth Cancer Institute-Anderson, Cincinnati, Ohio
  - Louis Stokes Cleveland VA Medical Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Mount Carmel East Hospital, Columbus, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Premier Blood and Cancer Center, Dayton, Ohio
  - Dayton Physician LLC - Englewood, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Dublin Methodist Hospital, Dublin, Ohio
  - Armes Family Cancer Center, Findlay, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Orion Cancer Care, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Dayton Physicians LLC-Atrium, Franklin, Ohio
  - Central Ohio Breast and Endocrine Surgery, Gahanna, Ohio
  - Dayton Physicians LLC-Wayne, Greenville, Ohio
  - Miami Valley Cancer Care and Infusion, Greenville, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Mount Carmel Grove City Hospital, Grove City, Ohio
  - Greater Dayton Cancer Center, Kettering, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Saint Rita's Medical Center, Lima, Ohio
  - OhioHealth Mansfield Hospital, Mansfield, Ohio
  - Cleveland Clinic Cancer Center Mansfield, Mansfield, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - OhioHealth Marion General Hospital, Marion, Ohio
  - Memorial Hospital, Marysville, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Newark Radiation Oncology, Newark, Ohio
  - Mercy Health - Perrysburg Hospital, Perrysburg, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - North Coast Cancer Care, Sandusky, Ohio
  - Springfield Regional Cancer Center, Springfield, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Trinity's Tony Teramana Cancer Center, Steubenville, Ohio
  - Cleveland Clinic Cancer Center Strongsville, Strongsville, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - Mercy Health - Saint Vincent Hospital, Toledo, Ohio
  - Mercy Health - Saint Anne Hospital, Toledo, Ohio
  - Dayton Physicians LLC - Troy, Troy, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Saint Joseph Warren Hospital, Warren, Ohio
  - South Pointe Hospital, Warrensville Heights, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Cleveland Clinic Wooster Family Health and Surgery Center, Wooster, Ohio
  - Saint Elizabeth Youngstown Hospital, Youngstown, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - Cancer Centers of Southwest Oklahoma Research, Lawton, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Saint Alphonsus Cancer Care Center-Baker City, Baker City, Oregon
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Cancer Institute Clackamas Clinic, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Saint Alphonsus Cancer Care Center-Ontario, Ontario, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Kaiser Permanente Northwest, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Saint Charles Health System-Redmond, Redmond, Oregon
  - Salem Hospital, Salem, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - UPMC Altoona, Altoona, Pennsylvania
  - UPMC-Heritage Valley Health System Beaver, Beaver, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - UPMC Hillman Cancer Center at Butler Health System, Butler, Pennsylvania
  - UPMC Camp Hill, Camp Hill, Pennsylvania
  - Carlisle Regional Cancer Center, Carlisle, Pennsylvania
  - Christiana Care Health System-Concord Health Center, Chadds Ford, Pennsylvania
  - Chambersburg Hospital, Chambersburg, Pennsylvania
  - WellSpan Medical Oncology and Hematology, Chambersburg, Pennsylvania
  - Fox Chase Cancer Center - East Norriton Hospital Outpatient Center, East Norriton, Pennsylvania
  - Pocono Medical Center, East Stroudsburg, Pennsylvania
  - Ephrata Cancer Center, Ephrata, Pennsylvania
  - Ephrata Community Hospital, Ephrata, Pennsylvania
  - UPMC Hillman Cancer Center Erie, Erie, Pennsylvania
  - UPMC Cancer Center at UPMC Horizon, Farrell, Pennsylvania
  - Adams Cancer Center, Gettysburg, Pennsylvania
  - UPMC Cancer Centers - Arnold Palmer Pavilion, Greensburg, Pennsylvania
  - UPMC Hillman Cancer Center in Greenville/UPMC Horizon, Greenville, Pennsylvania
  - WellSpan Medical Oncology and Hematology, Hanover, Pennsylvania
  - UPMC Pinnacle Cancer Center/Community Osteopathic Campus, Harrisburg, Pennsylvania
  - Lehigh Valley Hospital-Hazleton, Hazleton, Pennsylvania
  - IRMC Cancer Center, Indiana, Pennsylvania
  - UPMC-Johnstown/John P. Murtha Regional Cancer Center, Johnstown, Pennsylvania
  - Sechler Family Cancer Center, Lebanon, Pennsylvania
  - UPMC Cancer Center at UPMC McKeesport, McKeesport, Pennsylvania
  - UPMC Hillman Cancer Center at Rocco And Nancy Ortenzio Cancer Pavilion, Mechanicsburg, Pennsylvania
  - UPMC Hillman Cancer Center - Monroeville, Monroeville, Pennsylvania
  - UPMC Hillman Cancer Center in Coraopolis, Moon Township, Pennsylvania
  - UPMC Hillman Cancer Center - Part of Frick Hospital, Mount Pleasant, Pennsylvania
  - Arnold Palmer Cancer Center Medical Oncology Norwin, N. Huntingdon, Pennsylvania
  - UPMC Cancer Center-Natrona Heights, Natrona Heights, Pennsylvania
  - UPMC Hillman Cancer Center - New Castle, New Castle, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - UPMC-Saint Margaret, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - UPMC-Passavant Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Clair Hospital Cancer Center, Pittsburgh, Pennsylvania
  - Pottstown Hospital, Pottstown, Pennsylvania
  - UPMC Cancer Center at UPMC Northwest, Seneca, Pennsylvania
  - UPMC Cancer Center-Uniontown, Uniontown, Pennsylvania
  - UPMC Cancer Center-Washington, Washington, Pennsylvania
  - UPMC West Mifflin-Cancer Center Jefferson, West Mifflin, Pennsylvania
  - UPMC Susquehanna, Williamsport, Pennsylvania
  - Divine Providence Hospital, Williamsport, Pennsylvania
  - Cancer Care Associates of York, York, Pennsylvania
  - WellSpan Health-York Cancer Center, York, Pennsylvania
  - WellSpan Health-York Hospital, York, Pennsylvania
  - UPMC Memorial, York, Pennsylvania
  - Providence Veterans Administration Hospital, Providence, Rhode Island
  - Smilow Cancer Hospital Care Center - Westerly, Westerly, Rhode Island
  - AnMed Health Cancer Center, Anderson, South Carolina
  - Saint Joseph's/Candler - Bluffton Campus, Bluffton, South Carolina
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Ralph H Johnson VA Medical Center, Charleston, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Baptist Memorial Hospital and Cancer Center-Collierville, Collierville, Tennessee
  - Baptist Memorial Hospital and Cancer Center-Memphis, Memphis, Tennessee
  - The Don and Sybil Harrington Cancer Center, Amarillo, Texas
  - Saint Joseph Regional Cancer Center, Bryan, Texas
  - Parkland Memorial Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Fort Worth, Fort Worth, Texas
  - UT Southwestern Clinical Center at Richardson/Plano, Richardson, Texas
  - Central Vermont Medical Center/National Life Cancer Treatment, Berlin Corners, Vermont
  - University of Vermont Medical Center, Burlington, Vermont
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - White River Junction Veteran Administration Medical Center, White River Junction, Vermont
  - Kaiser Permanente-Burke Medical Center, Burke, Virginia
  - Centra Alan B Pearson Regional Cancer Center, Lynchburg, Virginia
  - Kaiser Permanente Tysons Corner Medical Center, McLean, Virginia
  - Bon Secours Memorial Regional Medical Center, Mechanicsville, Virginia
  - Bon Secours Westchester Emergency Center, Midlothian, Virginia
  - Bon Secours Saint Francis Medical Center, Midlothian, Virginia
  - Bon Secours DePaul Medical Center, Norfolk, Virginia
  - Bon Secours Maryview Medical Center, Portsmouth, Virginia
  - Bon Secours Saint Mary's Hospital, Richmond, Virginia
  - Virginia Cancer Institute, Richmond, Virginia
  - Bon Secours Cancer Institute at Reynolds Crossing, Richmond, Virginia
  - VCU Massey Cancer Center at Stony Point, Richmond, Virginia
  - Hunter Holmes McGuire Veterans Administration Medical Center, Richmond, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - VCU Community Memorial Health Center, South Hill, Virginia
  - Bon Secours Health Center at Harbour View, Suffolk, Virginia
  - Kaiser Permanente-Caton Hill Medical Center, Woodbridge, Virginia
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - Overlake Medical Center, Bellevue, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Saint Elizabeth Hospital, Enumclaw, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Jefferson Healthcare, Port Townsend, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - Valley Medical Center, Renton, Washington
  - Pacific Gynecology Specialists, Seattle, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Swedish Medical Center-Cherry Hill, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - PeaceHealth United General Medical Center, Sedro-Woolley, Washington
  - Providence Regional Cancer System-Shelton, Shelton, Washington
  - Saint Michael Cancer Center, Silverdale, Washington
  - Franciscan Research Center-Northwest Medical Plaza, Tacoma, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - Providence Regional Cancer System-Yelm, Yelm, Washington
  - Edwards Comprehensive Cancer Center, Huntington, West Virginia
  - Saint Mary's Medical Center, Huntington, West Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - Ascension Saint Elizabeth Hospital, Appleton, Wisconsin
  - Duluth Clinic Ashland, Ashland, Wisconsin
  - Northwest Wisconsin Cancer Center, Ashland, Wisconsin
  - Ascension Southeast Wisconsin Hospital - Elmbrook Campus, Brookfield, Wisconsin
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Ascension Calumet Hospital, Chilton, Wisconsin
  - Aurora Saint Luke's South Shore, Cudahy, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Ascension Saint Francis - Reiman Cancer Center, Franklin, Wisconsin
  - Ascension Southeast Wisconsin Hospital - Franklin, Franklin, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Aspirus Medford Hospital, Medford, Wisconsin
  - Ascension Columbia Saint Mary's Hospital Ozaukee, Mequon, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Ascension Southeast Wisconsin Hospital - Saint Joseph Campus, Milwaukee, Wisconsin
  - Ascension Columbia Saint Mary's Hospital - Milwaukee, Milwaukee, Wisconsin
  - Ascension Saint Francis Hospital, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - Ascension Mercy Hospital, Oshkosh, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Ascension All Saints Hospital, Racine, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Aspirus Cancer Care - James Beck Cancer Center, Rhinelander, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Aspirus Cancer Care - Stevens Point, Stevens Point, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Ascension Medical Group Southeast Wisconsin - Mayfair Road, Wauwatosa, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Aspirus Cancer Care - Wisconsin Rapids, Wisconsin Rapids, Wisconsin
  - Cheyenne Regional Medical Center-West, Cheyenne, Wyoming
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming
- FHP Health Center-Guam, Tamuning, Guam